CLINICAL TRIAL: NCT05190900
Title: Changes in Stabilometry After Neural Mobilisation of the Dorsocutaneous Lateral and Medial Posterior Tibial and Deep Peroneal Nerves.
Brief Title: Changes in Stabilometry After Neural Mobilisation in Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, PhD, principal investigator, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3010201915819 B
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Postural Balance; Foot; Therapy; Rehabilitation
Keywords: Platform; Stabilometry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): We will measure the stabilometric variables before and after the performance of a neuromeningeal mobilisation.
  Interventions: Other: neural mobilization

INTERVENTIONS:
Other: neural mobilization — neural mobilisation of the posterior tibial, deep peroneal and lateral, intermediate and medial dorsocutaneous nerves.

SUMMARY:
Investigation will consist of measuring before and after applying nerve mobilization exercise. Measurements will be made on the same day without the need to go at another time.

In this study, participants will be asked to stand on a pressure platform several times in a relaxed manner and with eyes open and closed before and after a neuromeningeal mobilization technique indicated for the treatment of pain in your feet. Measurements or tests to be carried out are totally innocuous and do not carry any risk to your health and integrity.

Participants will have to remain barefoot for a maximum of 30 seconds, a total of 8 times on a pressure platform

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed with active or latent MTrP in bilateral flexor digitorum brevis.
* MTrPs were the only MTrPs diagnosed in limb or foot.
* Participants had a normal body mass.
* Age range of 20 to 40 years.

Exclusion criteria:

* Diagnosis of lower limb injury.
* History of previous lower extremity surgery.
* Required not to have undergone ankle stretching or any other treatment
* Diabetes due to possible elevation of plantar pressure.
* Deformities of the toes, such as hammer toes and hallux valgus due to their possible alteration in plantar pressure.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Stabilometry variable x displacement open eyes before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with open eyes.
Stabilometry variable y displacement open eyes before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with open eyes.
Stabilometry variable center of pressure area open eyes before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes open.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction open eyes | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction open eyes before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with eyes closed.
Stabilometry variable y displacement before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with closed eyes.
Stabilometry variable center of pressure area before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes closed.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction before | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement open eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with open eyes.
Stabilometry variable y displacement open eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with open eyes.
Stabilometry variable center of pressure area open eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes open.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction with open eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction with open eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement with closed eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with eyes closed.
Stabilometry variable y displacement with closed eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with closed eyes.
Stabilometry variable center of pressure area with closed eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes closed.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction with closed eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction with closed eyes after intervention | Through study completion, an average of 2 days
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).

CONTACTS AND LOCATIONS:
Locations (1):
- EVA MARIA Martínez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There will be no plan to share

REFERENCES:
- [Derived] Martinez-Jimenez EM, Losa-Iglesias ME, Becerro-de-Bengoa-Vallejo R, Rodriguez-Sanz D, Calvo-Lobo C, Jimenez-Fernandez R, Corral-Liria I, Perez-Boal E, Navarro-Flores E. Effects of neural mobilization of sciatic nerve and its branches in plantar foot pressures and stabilometry. Sci Rep. 2024 Oct 8;14(1):23417. doi: 10.1038/s41598-024-72848-4. PMID 39379413